CLINICAL TRIAL: NCT04184622
Title: Efficacy and Safety of Tirzepatide Once Weekly in Participants Without Type 2 Diabetes Who Have Obesity or Are Overweight With Weight- Related Comorbidities: A Randomized, Double-Blind, Placebo-Controlled Trial (SURMOUNT-1)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight
Acronym: SURMOUNT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17244; I8F-MC-GPHK (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-12-02; First posted 2019-12-03 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Overweight; Obesity
Keywords: Metabolism and Nutrition Disorder; Prediabetes
MeSH Terms: conditions — Overweight; Obesity; Nutrition Disorders; Prediabetic State | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received once weekly (QW) subcutaneous (SC) doses of a matching placebo, administered over a period of 72 weeks.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the placebo dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
  Interventions: Drug: Placebo
- 5 mg Tirzepatide (Experimental): * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 milligrams (mg) and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 5 mg tirzepatide dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 10 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 10 mg tirzepatide dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 15 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 15 mg tirzepatide dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of tirzepatide in participants with overweight and obesity. The main purpose is to learn more about how tirzepatide affects body weight. The study has two phases: A main phase and an extension phase. The main phase of the study will last 72 weeks. Participants with prediabetes will continue in the extension for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Body mass Index (BMI) ≥30 kilograms per square meter (kg/m²), or ≥27 kg/m² and previous diagnosis with at least one of the following comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease
* History of at least one unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Diabetes mellitus
* Change in body weight greater than 5 kg within 3 months prior to starting study
* Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2539 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (118):
- United States (54):
  - Cahaba Research, Pelham, Alabama
  - Perseverance Research Center, Scottsdale, Arizona
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Research, Fresno, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Herman Clinical Research, Suwanee, Georgia
  - SKY Integrative Medical Center/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Premier Research, Trenton, New Jersey
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Detweiler Family Medicine & Associates, Lansdale, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
- Argentina (9):
  - Stat Research S.A., CABA, Buenos Aires
  - CEDIC, CABA, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - DIM Clinica Privada, Ramos Mejía, Buenos Aires
  - GO Centro Médico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
- Brazil (8):
  - CEDOES, Vitória, Espírito Santo
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Loema - Instituto de Pesquisa Clinica, Campinas, São Paulo
  - Instituto Brasil de Pesquisa Clínica - IBPCLIN, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital da Clinicas da Faculdade de Medicina da USP, São Paulo
- China (7):
  - Beijing Tsinghua Changgung Hospital, Changping, Beijing Municipality
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Ningbo First Hospital, Ningbo, Zhejiang
- India (6):
  - Gujarat Endocrine Center, Ahmedabad, Gujarat
  - Sir J.J. Group of Hospitals, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Care Hospitals Hyderabad- Banjara Hills, Hyderabad, Telangana
  - ILS Hospital, Kolkata, West Bengal
  - Fortis Hospital, Delhi
- Japan (5):
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - AMC Nishiumeda Clinic, Osaka
- Mexico (10):
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Unidad de Investigacion Clinica y Atencion Medica HEPA, Guadalajara, Jalisco
  - Virgen Cardiovascular Research S.C, Guadalajara, Jalisco
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - RM Pharma Specialists, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
  - Arké SMO S.A de C.V, Veracruz
- Puerto Rico (5):
  - Manati Center for Clinical Research, Manatí
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC- Hato Rey Site, San Juan
  - Private Practice - Dr. Luis Rivera Colon, San Juan
- Russia (9):
  - Ivanovo Regional Healthcare Institution Cardiology Dispensary, Ivanovo, Ivanovo Oblast
  - Immanuel Kant Baltic Federal University, Kaliningrad, Kaliningrad Oblast
  - Endocrinology Research Center of Rosmedtechnologies, Moscow, Moscow
  - Pirogov Russian National Research Medical University, Moscow, Moscow
  - Russian Cardiology Research and Production Complex, Moscow, Moscow
  - State Research Center for Preventive Medicine, Moscow, Moscow
  - Research Institute of Therapy and Preventive Medicine, Novosibirsk, Novosibirsk Oblast
  - St Petersburg SBHI City Hospital No. 38 Named After Semashko, Saint Petersburg, Sankt-Peterburg
  - Izhevsk City Clinical Hospital Number 9, Izhevsk, Udmurtiya Republic
- Taiwan (5):
  - Chi-Mei Medical Center, Tainan, Tainan
  - National Taiwan University Hospital, Taipei City, Taipei
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Ishigaki Y, Yamada M, Shingaki T, Oura T, Shimomura I. Efficacy and Safety of Tirzepatide in Japanese Participants With Obesity: A Subpopulation Analysis of the SURMOUNT-1 Trial. Obesity (Silver Spring). 2026 Jan 30. doi: 10.1002/oby.70131. Online ahead of print. PMID 41612966
- [Derived] Wadden TA, Oquendo MA, Kushner RF, Cao D, Karanikas CA, Kechter A, Murphy MA. Psychiatric Safety of Tirzepatide in People With Obesity and No Known Major Psychopathology: A Post Hoc Analysis of SURMOUNT. Obesity (Silver Spring). 2026 Jan 15. doi: 10.1002/oby.70122. Online ahead of print. PMID 41537305
- [Derived] Li X, Cao D, Sapin H, Wang F, Hunter Gibble T, Raibulet NK, Denning M, Kaplan LM. People With Lowest Physical Functioning Scores Showed Greatest Improvement After Tirzepatide Treatment. Obesity (Silver Spring). 2026 Jan;34(1):114-126. doi: 10.1002/oby.70067. Epub 2025 Nov 4. PMID 41187013
- [Derived] Gourgari E, Srivastava G, Kelly AS, Mojdami D, Cao D, Murphy MA, Karanikas CA, Lee CJ. Early-Onset Obesity and Tirzepatide Treatment: A Post Hoc Analysis of the SURMOUNT Clinical Trials. Obesity (Silver Spring). 2025 Sep;33(9):1668-1679. doi: 10.1002/oby.24348. Epub 2025 Jul 27. PMID 40717199
- [Derived] Ard J, Lee CJ, Gudzune K, Addison B, Lingvay I, Cao D, Mast CJ, Stefanski A, Falcon B, Mojdami D. Weight reduction over time in tirzepatide-treated participants by early weight loss response: Post hoc analysis in SURMOUNT-1. Diabetes Obes Metab. 2025 Sep;27(9):5064-5071. doi: 10.1111/dom.16554. Epub 2025 Jul 17. PMID 40677091
- [Derived] Linetzky B, Sattar N, Verma S, Krumholz HM, Xie CC, Hoffmann HT, Zimner-Rapuch S, Torcello-Gomez A, Stefanski A. Improvements in Cardiometabolic Risk Factors by Weight Reduction: A Post Hoc Analysis of Adults With Obesity Randomly Assigned to Tirzepatide. Ann Intern Med. 2025 Aug;178(8):1095-1105. doi: 10.7326/ANNALS-24-02623. Epub 2025 Jun 24. PMID 40550133
- [Derived] Heerspink HJL, Friedman AN, Bjornstad P, van Raalte DH, Cherney D, Cao D, Garcia-Perez LE, Stefanski A, Turfanda I, Bunck MC, Benabbad I, Griffin R, Piras de Oliveira C. Kidney Parameters with Tirzepatide in Obesity with or without Type 2 Diabetes. J Am Soc Nephrol. 2025 Nov 1;36(11):2190-2200. doi: 10.1681/ASN.0000000764. Epub 2025 Jun 13. PMID 40512543
- [Derived] Horn DB, Kahan S, Batterham RL, Cao D, Lee CJ, Murphy M, Gonsahn-Bollie S, Chigutsa F, Stefanski A, Dunn JP. Time to weight plateau with tirzepatide treatment in the SURMOUNT-1 and SURMOUNT-4 clinical trials. Clin Obes. 2025 Jun;15(3):e12734. doi: 10.1111/cob.12734. Epub 2025 Jan 12. PMID 39800653
- [Derived] Jastreboff AM, le Roux CW, Stefanski A, Aronne LJ, Halpern B, Wharton S, Wilding JPH, Perreault L, Zhang S, Battula R, Bunck MC, Ahmad NN, Jouravskaya I; SURMOUNT-1 Investigators. Tirzepatide for Obesity Treatment and Diabetes Prevention. N Engl J Med. 2025 Mar 6;392(10):958-971. doi: 10.1056/NEJMoa2410819. Epub 2024 Nov 13. PMID 39536238
- [Derived] Gudzune KA, Stefanski A, Cao D, Mojdami D, Wang F, Ahmad N, Ling Poon J. Association between weight reduction achieved with tirzepatide and quality of life in adults with obesity: Results from the SURMOUNT-1 study. Diabetes Obes Metab. 2025 Feb;27(2):539-550. doi: 10.1111/dom.16046. Epub 2024 Nov 4. PMID 39497468
- [Derived] Krumholz HM, de Lemos JA, Sattar N, Linetzky B, Sharma P, Mast CJ, Ahmad NN, Bunck MC, Stefanski A. Tirzepatide and blood pressure reduction: stratified analyses of the SURMOUNT-1 randomised controlled trial. Heart. 2024 Sep 16;110(19):1165-1171. doi: 10.1136/heartjnl-2024-324170. PMID 39084707
- [Derived] Hankosky ER, Wang H, Neff LM, Kan H, Wang F, Ahmad NN, Stefanski A, Garvey WT. Tirzepatide reduces the predicted risk of developing type 2 diabetes in people with obesity or overweight: Post hoc analysis of the SURMOUNT-1 trial. Diabetes Obes Metab. 2023 Dec;25(12):3748-3756. doi: 10.1111/dom.15269. Epub 2023 Sep 12. PMID 37700443
- [Derived] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- See also: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight — https://trials.lillytrialguide.com/en-US/trial/1o8ZY82Yn01Z4Hqvx0WuME

RESULTS

PARTICIPANT FLOW:
Period: Primary Treatment Period
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Started (Participants with normoglycemia or prediabetes at the time of randomization were eligible to enter this primary treatment period.) | 643 | 630 | 636 | 630
Received at Least One Dose of Study Drug | 643 | 630 | 636 | 630
Participants With Normoglycemia at Randomization | 373 | 383 | 374 | 377
Participants With Prediabetes at Randomization | 270 | 247 | 262 | 253
Completed | 509 | 569 | 566 | 575
Not Completed | 134 | 61 | 70 | 55
Not completed — Adverse Event | 6 | 4 | 8 | 6
Not completed — Death | 4 | 4 | 2 | 1
Not completed — Lost to Follow-up | 41 | 17 | 15 | 13
Not completed — Other - as reported by the investigator | 21 | 7 | 6 | 12
Not completed — Physician Decision | 0 | 0 | 3 | 1
Not completed — Pregnancy | 4 | 3 | 4 | 1
Not completed — Withdrawal by Subject | 58 | 26 | 32 | 21
Period: Additional Treatment Period
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Started (Only participants from the primary treatment period who had prediabetes at the time of randomization were eligible to enter the additional treatment period.) | 213 | 227 | 229 | 232
Completed | 182 | 201 | 211 | 217
Not Completed | 31 | 26 | 18 | 15
Not completed — Adverse Event | 1 | 2 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 6 | 4 | 8 | 6
Not completed — Other - as reported by the investigator | 2 | 5 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Not completed — Site closed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 21 | 15 | 3 | 7
Period: Safety Follow-up Period
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Started (Participants who completed or discontinued either the primary or additional treatment periods entered the safety follow-up period.) | 478 | 543 | 548 | 560
Entered From Primary Treatment Period | 328 | 362 | 355 | 367
Entered From Additional Treatment Period | 150 | 181 | 193 | 193
Completed | 421 | 508 | 514 | 518
Not Completed | 57 | 35 | 34 | 42
Not completed — Adverse Event | 6 | 8 | 9 | 16
Not completed — Lost to Follow-up | 4 | 4 | 10 | 3
Not completed — Missing Weight at Week 176 | 3 | 2 | 2 | 2
Not completed — Other - as reported by the investigator | 10 | 5 | 6 | 5
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 3 | 0 | 6
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 31 | 13 | 7 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Placebo: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of a matching placebo, administered over a period of 72 weeks.
- 5 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg, which was then maintained up to week 72.
- 10 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 10 mg, which was then maintained up to week 72.
- 15 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 15 mg, which was then maintained up to week 72.
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Total
Number analyzed (Participants) | 643 | 630 | 636 | 630 | 2539
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.5) | 45.6 (12.7) | 44.7 (12.4) | 44.9 (12.3) | 44.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436 | 426 | 427 | 425 | 1714
  Male | 207 | 204 | 209 | 205 | 825
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 58 | 56 | 58 | 59 | 231
  Asian | 71 | 68 | 71 | 66 | 276
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 2 | 3 | 9
  Black or African American | 55 | 48 | 47 | 51 | 201
  White | 450 | 447 | 452 | 443 | 1792
  More than one race | 7 | 9 | 6 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 93 | 90 | 90 | 91 | 364
  United States | 288 | 282 | 287 | 284 | 1141
  Japan | 33 | 30 | 30 | 31 | 124
  China | 7 | 9 | 7 | 7 | 30
  Taiwan | 15 | 12 | 15 | 16 | 58
  Brazil | 59 | 59 | 61 | 60 | 239
  Mexico | 108 | 110 | 107 | 108 | 433
  Russia | 32 | 29 | 30 | 27 | 118
  India | 8 | 9 | 9 | 6 | 32
Baseline Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 104.9 (21.37) | 102.88 (20.71) | 105.84 (23.32) | 105.59 (22.92) | 104.78 (22.12)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight (Primary Treatment Period)
Description: Least Squares (LS) Mean was calculated using mixed-model repeated measures (MMRM) with baseline, analysis country, sex, prediabetes status at randomization, treatment, time, treatment*time (Type III sum of squares) in the model.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline body weight value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
percent change | -2.4 (0.40) | -16.0 (0.39) | -21.4 (0.39) | -22.5 (0.39)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Square (LS) Mean Difference (Net) = -13.5, 95% CI 2-sided [-14.6 to -12.5]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -18.9, 95% CI 2-sided [-20.0 to -17.8]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -20.1, 95% CI 2-sided [-21.2 to -19.0]

2. Primary Outcome: Percentage of Participants Who Achieve ≥5% Body Weight Reduction (Primary Treatment Period)
Description: Percentage of participants who achieve greater than or equal to( ≥) 5% body weight reduction.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥5% Body Weight Reduction, excluding data after prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
Percentage of Participants | 27.87 | 89.41 | 96.18 | 96.32
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 23.99, 95% CI 2-sided [17.43 to 33.02]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 73.63, 95% CI 2-sided [46.98 to 115.39]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 75.48, 95% CI 2-sided [47.86 to 119.03]

3. Secondary Outcome: Change From Baseline in Body Weight (Pooled Doses of Tirzepatide 10 mg and 15 mg) - Primary Treatment Period
Description: LS Mean was calculated using MMRM with baseline, analysis country, sex, prediabetes status at randomization, treatment, time, treatment*time (Type III sum of squares) in the model.
Time Frame: Baseline, Week 20
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline body weight value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 10 mg and 15 mg tirzepatide.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Groups:
- Pooled 10 mg/15 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 10 mg or 15mg, which was then maintained up to week 72.
Arm/Group | Placebo | Pooled 10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 635 | 1254
kilograms | -2.5 (0.22) | -13.2 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -10.7, 95% CI 2-sided [-11.2 to -10.1]

4. Secondary Outcome: Percentage of Participants Who Achieve ≥10% Body Weight Reduction (Primary Treatment Period)
Description: Percentage of Participants who Achieve ≥10% Body Weight Reduction
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥10% Body Weight Reduction, excluding data after prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
Percentage of Participants | 13.54 | 73.35 | 85.85 | 90.08
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 19.03, 95% CI 2-sided [14.15 to 25.60]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 44.17, 95% CI 2-sided [31.75 to 61.45]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 65.64, 95% CI 2-sided [45.94 to 93.77]

5. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction (Primary Treatment Period)
Description: Percentage of participants who achieve ≥15% body weight reduction.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥15% body weight reduction, excluding data after prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
Percentage of Participants | 5.98 | 50.24 | 73.61 | 78.24
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.08, 95% CI 2-sided [11.83 to 24.66]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 51.84, 95% CI 2-sided [35.42 to 75.88]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 66.63, 95% CI 2-sided [45.23 to 98.16]

6. Secondary Outcome: Percentage of Participants Who Achieve ≥20% Body Weight Reduction (Primary Treatment Period)
Description: Percentage of participants who achieve ≥20% body weight reduction.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥20% Body Weight Reduction, excluding data after prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
Percentage of Participants | 1.26 | 31.62 | 55.48 | 62.88
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 36.93, 95% CI 2-sided [18.37 to 74.22]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 109.45, 95% CI 2-sided [54.50 to 219.81]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 150.59, 95% CI 2-sided [74.85 to 302.97]

7. Secondary Outcome: Change From Baseline in Waist Circumference (Primary Treatment Period)
Description: as for outcome 3
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline weight circumference value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 634 | 622 | 629 | 625
centimeters | -3.4 (0.42) | -14.6 (0.41) | -19.4 (0.41) | -19.9 (0.41)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -11.2, 95% CI 2-sided [-12.3 to -10.0]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -16.0, 95% CI 2-sided [-17.2 to -14.9]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -16.5, 95% CI 2-sided [-17.7 to -15.4]

8. Secondary Outcome: Change From Baseline in Short Form Survey-36 Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score at Week 72 (Pooled Doses of Tirzepatide 10 mg and 15 mg) - Primary Treatment Period
Description: The SF-36v2 acute, 1-week recall version is a 36-item, generic, patient-administered measure designed to assess the following 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" while the remaining domains assess functioning "in the past week." Each domain is scored individually and information from these 8 domains are further aggregated into 2 health-component summary scores: Physical-Component Summary and Mental-Component Summary. Items are answered on Likert scales of varying lengths (3-, 5-, or 6- point scales).The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline SF-36v2 value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 10 mg and 15 mg tirzepatide.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pooled 10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 482 | 1080
score on a scale | 1.7 (0.27) | 4.0 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Net) = 2.3, 95% CI 2-sided [1.6 to 2.9]

9. Secondary Outcome: Percent Change From Baseline in Triglycerides (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Percent change from baseline in triglycerides are reported as model-based estimate and Standard Error (SE) from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had a baseline and at least one post-baseline triglyceride value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Pooled 5 mg/10 mg/15 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5mg,10 mg or 15mg, which was then maintained up to week 72.
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 612 | 1822
percent change | -6.3 (1.55) | -27.6 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -22.7, 95% CI 2-sided [-25.6 to -19.8]

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Results are reported as model-based estimate and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline total cholesterol value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Pooled 5 mg/10 mg/15 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg, 10 mg or 15 mg, which was then maintained up to week 72.
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 612 | 1822
percent change | -1.11 (0.695) | -5.97 (0.364)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -4.91, 95% CI 2-sided [-6.40 to -3.41]

11. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein (HDL) Cholesterol at Week 72 (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Results are reported as model-based estimate and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline total cholesterol HDL value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 581 | 1764
percent change | 0.25 (0.757) | 7.92 (0.447)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = 7.65, 95% CI 2-sided [5.85 to 9.49]

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline SBP value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 634 | 1878
millimeter of mercury (mmHg) | -1.3 (0.48) | -8.1 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -6.8, 95% CI 2-sided [-7.9 to -5.7]

13. Secondary Outcome: Percent Change From Baseline in Fasting Insulin (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Fasting Insulin is a test used to measure the amount of insulin in the body. Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had a baseline and at least one post-baseline fasting insulin value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 590 | 1779
percent change | -9.7 (2.60) | -46.9 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -41.2, 95% CI 2-sided [-44.9 to -37.3]

14. Secondary Outcome: Percent Change From Baseline in Body Weight (Primary and Additional Treatment Periods : Participants With Prediabetes at Randomization)
Description: LS Mean was calculated using mixed-model repeated measures (MMRM) with baseline, analysis country, sex, treatment, time, treatment*time (Type III sum of squares) in the model.
Time Frame: Baseline, Week 176
Population: Participants with prediabetes at randomization who received at least one dose of study drug and had baseline and at least one post-baseline body weight value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of a matching placebo, administered over a period of 72 weeks.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the placebo dose SC QW until week 176.
- 5 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 5 mg tirzepatide dose SC QW until week 176.
- 10 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 10 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 10 mg tirzepatide dose SC QW until week 176.
- 15 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 15 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 15 mg tirzepatide dose SC QW until week 176.
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 264 | 245 | 260 | 249
percent change | -2.1 (0.78) | -15.4 (0.74) | -19.9 (0.72) | -22.9 (0.73)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference (Net) = -13.2, 95% CI 2-sided [-15.3 to -11.1]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference (Net) = -17.7, 95% CI 2-sided [-19.8 to -15.7]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference (Net) = -20.7, 95% CI 2-sided [-22.8 to -18.6]

15. Secondary Outcome: Percentage of Participants With Onset of Type 2 Diabetes From Baseline to Week 176 (Primary and Additional Treatment Periods: Participants With Prediabetes at Randomization)
Description: The percentage of participants with onset of Type 2 diabetes mellitus (T2DM), evaluated as time to onset of T2DM among those who had pre-diabetes at randomization, was reported.
  Time to onset of Type 2 diabetes mellitus was defined as the duration from the date of randomization to the adjudication committee-confirmed date of incident diabetes. Participants who did not experience the event were censored.
Time Frame: Baseline through Week 176
Population: Participants with prediabetes at randomization who received at least one dose of study drug (including the censored participants). Number of participants censored in Placebo = 236, Pooled 5 mg/10 mg/15 mg Tirzepatide = 753.
Measure: Number; unit: Percentage of Participants
Groups:
- Pooled 5 mg/10 mg/15 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5mg,10 mg or 15mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 5mg,10 mg or 15mg, tirzepatide dose SC QW until week 176.
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 270 | 762
Percentage of Participants | 12.6 | 1.2
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.06, 95% CI 2-sided [0.03 to 0.13]

16. Secondary Outcome: Percentage of Participants With Onset of Type 2 Diabetes From Baseline to Week 193 (Primary and Additional Treatment Periods + Safety Follow-up Period: Participants With Prediabetes at Randomization)
Description: as for outcome 15
Time Frame: Baseline through Week 193
Population: Participants with prediabetes at randomization who received at least one dose of study drug (including the censored participants). Number of participants censored in Placebo = 233, Pooled 5 mg/10 mg/15 mg Tirzepatide = 744.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of a matching placebo, administered over a period of 72 weeks.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the placebo dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193).
- Pooled 5 mg/10 mg/15 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5mg,10 mg or 15mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 5mg,10 mg or 15mg, tirzepatide dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193).
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 270 | 762
Percentage of Participants | 13.7 | 2.4
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.07 to 0.21]

17. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) - Primary Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline BMI value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 635 | 623 | 629 | 625
kilograms per meter squared (kg/m^2) | -0.9 (0.16) | -5.9 (0.16) | -8.1 (0.16) | -8.6 (0.16)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -5.1, 95% CI 2-sided [-5.5 to -4.6]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -7.2, 95% CI 2-sided [-7.7 to -6.8]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -7.7, 95% CI 2-sided [-8.2 to -7.3]

18. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) - Primary Treatment Period
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS Mean was calculated using MMRM with baseline, analysis country, sex, prediabetes status at randomization, treatment, time, treatment*time (Type III sum of squares) in the model.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline HbA1c value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 612 | 607 | 607 | 608
Percentage of HbA1c | -0.07 (0.012) | -0.40 (0.012) | -0.49 (0.012) | -0.51 (0.012)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.36 to -0.30]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.45 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.48 to -0.41]

19. Secondary Outcome: Change From Baseline in Fasting Glucose (Primary Treatment Period)
Description: as for outcome 3
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline fasting glucose value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 612 | 608 | 606 | 608
milligram per deciliter (mg/dL) | 0.86 (0.514) | -7.73 (0.484) | -9.73 (0.486) | -10.55 (0.486)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -8.59, 95% CI 2-sided [-9.97 to -7.20]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -10.59, 95% CI 2-sided [-11.98 to -9.21]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -11.42, 95% CI 2-sided [-12.80 to -10.30]

20. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein (LDL) Cholesterol (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Results are reported as model-based estimate and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had a baseline and at least one post-baseline LDL value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Pooled 5 mg/10 mg/15 mg Tirzepatide: Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg,10 mg or 15 mg, which was then maintained up to week 72.
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 578 | 1754
percent change | -0.85 (1.076) | -6.86 (0.555)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -6.06, 95% CI 2-sided [-8.32 to -3.75]

21. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein (VLDL) Cholesterol (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Results are reported as model-based estimate and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline VLDL value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 577 | 1754
percent change | -5.6 (1.55) | -27.6 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -23.3, 95% CI 2-sided [-26.1 to -20.4]

22. Secondary Outcome: Percent Change From Baseline in Free Fatty Acids (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: Results are reported as model-based estimate and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline free fatty acids value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 576 | 1756
percent change | 6.1 (2.65) | -5.9 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -11.3, 95% CI 2-sided [-16.1 to -6.2]

23. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg) - Primary Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline DBP value, excluding data after prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Pooled 5 mg/10 mg/15 mg Tirzepatide
Number analyzed (Participants) | 634 | 1878
mmHg | -1.0 (0.35) | -5.3 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Pooled 5 mg/10 mg/15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Net) = -4.2, 95% CI 2-sided [-5.0 to -3.5]

24. Secondary Outcome: Percentage of Participants Who Achieve ≥5% Body Weight Reduction (Primary and Additional Treatment Periods : Participants With Prediabetes at Randomization)
Description: Percentage of Participants Who Achieve ≥5% Body Weight Reduction.
Time Frame: Week 176
Population: Participants with prediabetes at randomization who received at least one dose of study drug and had baseline and at least one post-baseline value for body weight, excluding data after prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 264 | 245 | 260 | 249
Percentage of Participants | 24.62 | 90.61 | 91.92 | 94.78
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 29.79, 95% CI 2-sided [17.73 to 50.05]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 35.05, 95% CI 2-sided [20.63 to 59.53]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 55.05, 95% CI 2-sided [29.61 to 102.34]

25. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite-Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score at Week 72 (Primary Treatment Period)
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific patient-reported outcomes (PRO) instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items), and psychosocial (13 items). A 5-item subset of the physical domain, the physical-function composite is also supported. Items in the physical-function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline IWQOL-Lite CT value, excluding data after prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 477 | 545 | 539 | 535
score on a scale | 10.1 (0.78) | 17.8 (0.73) | 20.7 (0.73) | 21.8 (0.73)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Net) = 7.7, 95% CI 2-sided [5.6 to 9.8]
Statistical Analysis 2: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Net) = 10.7, 95% CI 2-sided [8.6 to 12.8]
Statistical Analysis 3: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Net) = 11.7, 95% CI 2-sided [9.6 to 13.8]

26. Secondary Outcome: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Tirzepatide (Primary Treatment Period)
Description: PK: Steady State AUC of Tirzepatide. each participant will be assigned via the Interactive Web Response System (IWRS) to one of the sampling PK time windows of 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours postdose.
Time Frame: Week 8, 16, and 36, at 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours postdose
Population: All randomly assigned participants who are exposed to at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 626 | 629 | 625
nanograms*hours per milliliter (ng*h/mL) | 88900 (20.2) | 177000 (22.0) | 266000 (20.4)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 193
Description: * All randomized participants who received at least 1 dose of the study drug.
  * As per the pre-specified statistical analysis plan, safety data were analyzed and reported by randomized arms regardless of the actual treatment received by the participant.
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of a matching placebo, administered over a period of 72 weeks.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the placebo dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
- 5 mg Tirzepatide: * Primary Treatment Period (Week 0-Week 72): Participants with normoglycemia or prediabetes at the time of randomization received QW SC doses of tirzepatide, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks until reaching a dose of 5 mg, which was then maintained up to week 72.
  * Additional Treatment Period (Week 72-Week 176): At week 72, only participants who had prediabetes at the time of randomization and had completed the primary treatment period continued receiving the 5 mg tirzepatide dose SC QW until week 176.
  * Safety Follow-up Period: Participants who had completed or discontinued the primary treatment period were followed for safety for 4 weeks (weeks 72 - week 76), and those who had completed or discontinued the additional treatment period (prediabetes at randomization) were followed for 17 weeks (week 176 - week 193). No treatment was administered during this period.
Arm/Group | Placebo | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 4/643 | 4/630 | 3/636 | 2/630
Serious Adverse Events (participants affected / at risk) | 53/643 | 57/630 | 60/636 | 50/630
Other Adverse Events (participants affected / at risk) | 315/643 | 443/630 | 451/636 | 429/630
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=643) | 5 mg Tirzepatide (N=630) | 10 mg Tirzepatide (N=636) | 15 mg Tirzepatide (N=630)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear canal stenosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 3 (3) | 6 (6) | 7 (7)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sphincter of oddi dysfunction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 6 (6) | 2 (2) | 5 (5) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 4 (4) | 7 (7) | 4 (4) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0/436 (0) | 0/426 (0) | 0/427 (0) | 1/425 (1)
Peritoneal tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Central cord syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/436 (1) | 0/426 (0) | 0/427 (0) | 0/425 (0)
Adenosquamous carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/436 (0) | 0/426 (0) | 0/427 (0) | 1/425 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/436 (0) | 1/426 (1) | 0/427 (0) | 0/425 (0)
Gallbladder cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/436 (0) | 1/426 (1) | 0/427 (0) | 0/425 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/436 (1) | 0/426 (0) | 0/427 (0) | 0/425 (0)
Ovarian germ cell endodermal sinus tumour stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/436 (0) | 1/426 (1) | 0/427 (0) | 0/425 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/207 (0) | 1/204 (1) | 0/209 (0) | 0/205 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/207 (1) | 0/204 (0) | 0/209 (0) | 0/205 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/436 (0) | 0/426 (0) | 0/427 (0) | 2/425 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Idiopathic generalised epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/436 (0) | 1/426 (1) | 0/427 (0) | 0/425 (0)
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0/436 (0) | 1/426 (1) | 0/427 (0) | 0/425 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0/436 (0) | 0/426 (0) | 0/427 (0) | 1/425 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 0/436 (0) | 0/426 (0) | 0/427 (0) | 1/425 (1)
Cystocele (Reproductive system and breast disorders) | 0/436 (0) | 0/426 (0) | 1/427 (1) | 0/425 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/436 (0) | 0/426 (0) | 1/427 (1) | 0/425 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine fibrosis (Reproductive system and breast disorders) | 0/436 (0) | 0/426 (0) | 1/427 (1) | 0/425 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0/436 (0) | 0/426 (0) | 1/427 (1) | 0/425 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/436 (1) | 0/426 (0) | 0/427 (0) | 0/425 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Homicide (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=643) | 5 mg Tirzepatide (N=630) | 10 mg Tirzepatide (N=636) | 15 mg Tirzepatide (N=630)
Abdominal pain (Gastrointestinal disorders) | 24 (28) | 38 (52) | 38 (56) | 33 (62)
Constipation (Gastrointestinal disorders) | 38 (49) | 113 (129) | 117 (148) | 80 (100)
Diarrhoea (Gastrointestinal disorders) | 51 (90) | 128 (209) | 143 (281) | 149 (326)
Dyspepsia (Gastrointestinal disorders) | 31 (34) | 59 (88) | 64 (82) | 74 (126)
Eructation (Gastrointestinal disorders) | 4 (4) | 24 (32) | 35 (37) | 35 (159)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (17) | 31 (35) | 28 (29) | 34 (41)
Nausea (Gastrointestinal disorders) | 63 (103) | 160 (404) | 217 (540) | 201 (506)
Vomiting (Gastrointestinal disorders) | 12 (13) | 58 (82) | 74 (122) | 81 (144)
Injection site reaction (General disorders) | 2 (2) | 18 (175) | 36 (229) | 29 (223)
Covid-19 (Infections and infestations) | 106 (117) | 127 (137) | 128 (141) | 113 (125)
Upper respiratory tract infection (Infections and infestations) | 30 (36) | 32 (39) | 30 (46) | 30 (44)
Urinary tract infection (Infections and infestations) | 38 (47) | 30 (37) | 38 (42) | 28 (28)
Decreased appetite (Metabolism and nutrition disorders) | 22 (25) | 60 (65) | 75 (87) | 55 (72)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 36 (36) | 5 (5) | 9 (9) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (24) | 32 (33) | 20 (28) | 25 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (29) | 31 (36) | 30 (34) | 34 (35)
Dizziness (Nervous system disorders) | 16 (17) | 31 (36) | 37 (46) | 27 (34)
Headache (Nervous system disorders) | 47 (53) | 47 (57) | 51 (69) | 44 (56)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 33 (35) | 32 (33) | 37 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04184622/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT04184622/SAP_001.pdf